CLINICAL TRIAL: NCT04729335
Title: Detection and Application of Organic Disease With Phonocardiac Spectrometry
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-Shun Wu, Dr., Taipei Medical University WanFang Hospital
Other Study IDs: N201805104
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Phonocardiography
Keywords: phonocardiac spectrometry, organic disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: phonocardiac spectrometry — Detection and application of organic disease with phonocardiac spectrometry

SUMMARY:
Western medicine, as to disease detection, is based on histological pathology and organ anatomy, therefore biochemistry and medical imageology were developed to determine the location and mechanism of the sickness. Chinese medicine, in the other way around, follow the harmony between man and nature, creating four ways of diagnosis, namely looking, listening, questioning and pulse feeling, which evaluate the physiological homeostasis by the yin-yang of qi and blood, further judging the energy exchange between individual and the universe.

DETAILED DESCRIPTION:
Western medicine, as to disease detection, is based on histological pathology and organ anatomy, therefore biochemistry and medical imageology were developed to determine the location and mechanism of the sickness. Chinese medicine, in the other way around, follow the harmony between man and nature, creating four ways of diagnosis, namely looking, listening, questioning and pulse feeling, which evaluate the physiological homeostasis by the yin-yang of qi and blood, further judging the energy exchange between individual and the universe.

Pulse sound provides perfect detection of disease in Chinese medicine. Hence we plan to digitalize the pulse sound for a better interpretation of the sickness. According to past studies of pulse sound from radial artery, the lower frequency is below 25Hz, which falls into the detection range of Messener's corpuscles (2-80Hz), which are located intensively in index and middle fingers. However, radial artery is relative thinner and the pulse sound is not easy to target by the microphone, not to mention the interference from artery sclerosis. To this end our research group developed Phonocardiac spectrometry (PCS) to replace the traditional pulse instrument.

Since heart beats continuously, we hypothesize that each organ is regularly sending the signal back to heart, which modulate the contraction and beating of heart, reflecting different state of each organ. Heart is just like the commander of an orchestra band, who can direct the rhythm and style of the band by the music score and instruments. Once the instrument is damaged, the commander (heart) also adjusts himself. PCS can easily locate the pulse sound, and directly detect and analyze the cardiac spectrum. The real-time state in heart-organ axis can be readily monitored, recorded and investigated by PCS.

Our preliminary analysis focuses on patients with liver and pancreatic cancers. The results demonstrate the different pattern of cardiac spectrum between patients and normal people, which can be further sorted by disease types. By applying PCS measurement and the novel algorithm calculation to various diseases, we aim to build up a novel platform for disease screening or even diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer, out- and in-patients in gastroenterology division of Wanfang hospital.

Exclusion Criteria:

* 1.The decline and fall of informed consent.
* 2.Pregnancy.
* 3.Heart murmur grading greater or equal to level 3.
* 4.Cardiac Arrhythmia.
* 5.Patient with critical conditions such as renal or heart failure.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer, out- and in-patients in gastroenterology division of Wanfang hospital.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Readout of phonocardiac spectrometry for organ disease | 6 months
  Readout of phonocardiac spectrometry for organ disease

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shun Wu, Study Director — Taipei Municipal Wanfang Hospital
Locations (1):
- Wanfang Hospital, Taipei, Wenshan District, Taiwan

IPD SHARING:
Plan to Share IPD: No